CLINICAL TRIAL: NCT04915144
Title: A Prospective Randomized Study of the Efficacy and Safety of 177Lu-DOTATOC With Either Standard or Personalized Dosing for the Treatment of Patients With Somatostatin Receptor Positive NETs
Brief Title: 177Lu-DOTATOC for the Treatment of Patients With Somatostatin Receptor Positive NETs
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator decision
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H20-03401
Record Dates: First submitted 2021-04-28; First posted 2021-06-07 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Neuroendocrine Tumors; Carcinoid Tumor; Pulmonary Carcinoid Tumor; Gastroenteropancreatic Neuroendocrine Tumor; Vipoma; Insulinoma; Gastrinoma
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor; Gastro-enteropancreatic neuroendocrine tumor; Vipoma; Insulinoma; Gastrinoma | interventions — 177Lu-octreotide, DOTA(0)-Tyr(3)-

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized phase II study two-arm study of efficacy and safety of 177Lu-DOTATOC for treatment of patients with NETs who are referred to BC Cancer - Vancouver for treatment of progressive tumours.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard PRRT (Active Comparator): For standard PRRT 177Lu-DOTATOC therapy, the administered activity will be 7.4 GBq ± 10% as an intravenous infusion over a time of 10 to 30 minutes.
  Interventions: Drug: 177Lu-DOTATOC
- Personalized PRRT (Experimental): For 177Lu-DOTATOC therapy, for the first cycle the administered activity will be 7.4 GBq ± 10% as an intravenous infusion over a time of 10 to 30 minutes.Subsequent cycles will be adjusted based on dosimetry calculations.
  Interventions: Drug: 177Lu-DOTATOC

INTERVENTIONS:
Drug: 177Lu-DOTATOC — Subjects will receive 177Lu-DOTATOC PRRT treatment over 4 cycles, each cycle occurs every 8 weeks.

SUMMARY:
This study is to assess if personalized peptide receptor radionuclide therapy (PRRT) with 177Lu-DOTATOC results in fewer adverse events than standard PRRT. Subjects will be randomized to either receive personalized or standard PRRT. Personalized PRRT will be determined based on dosimetry calculations after the first cycle. In addition comparisons, will be made with progression-free survival, serial CT imaging, ctDNA, and quality of life questionnaires. Subjects will be followed for 5 years or until they have progression and are switched to another systemic treatment (not including treatment with somatostatin analogues).

DETAILED DESCRIPTION:
Overall, 200 subjects will be randomized (1:1 randomization ratio) to receive standard injected activities of 177Lu-DOTATOC PRRT or personalized injection of 177Lu-DOTATOC PRRT. Randomization will be stratified for grade and primary location.

Screening Phase: Subjects will be screened against the inclusion and exclusion criteria. Screening by SSR imaging will be completed to determine expression of SSR and feasibility of treatment by PRRT. Once eligibility has been confirmed they will be randomized. Subjects will undergo a physical exam, complete a medical history questionnaire, quality of life questionnaires, blood work, and a diagnostic CT.

Treatment Phase: During the treatment phase, subjects will undergo 4 cycles of treatment. Each treatment cycle will be followed by 2 dosimetry SPECT/CT scans on day 1 (18 - 32 hours after treatment administration) and day 2 (64 - 80h after treatment administration) After cycle 3 quality of life questionnaires will be completed again.

Follow up Phase: At the end of treatment or after discontinuation of any cause, subjects will be followed for 5 years to continue data collection for the other objectives. Objective tumour response will be assessed every 6 months by diagnostic CT according to the RECIST 1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Age greater than or equal to 19 years
* Biopsy-proven, well-differentiated grade 1 - 3 NET
* Gastroenteropancreatic tumors (e.g. carcinoids, gastrinoma, insulinoma, glucagonoma, VIPoma, etc.), functioning and non-functioning
* Sympathoadrenal system tumors (phaeochromocytoma, paraganglioma)
* Pulmonary NET, functioning and non-functioning
* Easter Cooperative Oncology Group (ECOG) ≤ 2
* Ki67 ≤ 55%
* Progressive disease demonstrated by RECIST 1.1 criteria within the 6 months preceding the study.
* Patients with other evidence of progressive disease that is not demonstrated on CT (like rising biomarkers) may be included, at the discretion of the Tumour Review Board.
* If response to other treatments is considered adequate according to other criteria, the Tumour Review Board may consider excluding the patient from participation in the study.
* Tumour Review Board confirmation of suitability to proceed to PRRT treatment and enrollment in this trial.
* Positive PET SSR imaging (Krenning score 2 or higher) in previous 6 months (68Ga-DOTATOC, 68Ga-DOTATATE, 18F-AmBF3-TATE). If PET SSR imaging is not available 111In-penetreotide scintigraphy (Octreotide scan) is acceptable.
* Adequate laboratory parameters within two weeks of enrollment
* Kidneys

  * Serum creatinine ≤ 150 µmol/L
  * GFR ≥ 40 ml/min (using plasma clearance values)
* Marrow

  * Hemoglobin ≥ 80 g/L
  * WBC ≥ 2 x 109/L
  * Platelets ≥ 75 x 109/L
  * Liver
* Total bilirubin ≤ 3 x upper limit of normal (ULN)
* ALT ≤ 3 x ULN or ≤ 5 x ULN if liver metastasis
* Alkaline phosphatase ≤ 3 x ULN or ≤ 5 x ULN if liver metastasis
* Subject's ability to comply with scheduled visits, treatment plans, laboratory tests, imaging tests, and other procedures required as detailed in the protocol.

Exclusion Criteria:

* Women and men of childbearing potential Procreation

  * Women: pregnancy test done before enrollment before each treatment cycle. And subject must use adequate contraception for the duration of therapy, be surgically sterile, or post-menopausal.
  * Men: must be surgically sterile or use adequate contraception for the duration of the therapy.
* Patient with another non-cutaneous (excluding melanoma) active cancer requiring therapeutic intervention.
* Curative medical or surgical treatment, local liver embolization, or debulking are appropriate options.
* Life expectancy is less than 12 weeks.
* Radiotherapy to target lesions ≤ 12 weeks ago or to more than 25% of bone marrow.
* PRRT at any time prior to randomization in this study.
* Systemic therapy (chemotherapy) within 4 weeks of PRRT and other locoregional therapies (radioisotope, embolization) within 12 weeks prior to enrollment. Ongoing use of somatostatin analogs for control of symptoms is allowed.
* Known brain metastases (unless treated and stable for more than 3 months).
* Co-morbidities that could, in the opinion of the PI, interfere with safe delivery of PRRT (like urinary incontinence, psychiatric illness), uncontrolled congestive heart failure (NYHA II, III, IV)
* Breastfeeding (if patients elect to discontinue breast feeding, they can participate in the trial).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine whether personalized 177Lu-DOTATOC PRRT reduces adverse events (AE). | 8 months
  Frequency of AEs, will be compared between the two treatment arms.
Compare the 12-month progression-free survival (PFS) of subjects receiving personalized or standard injected activity PRRT with RECIST criteria. | 12 months
  PFS will be determined by RECIST1.1 criteria on serial CT, and analysed independently. The 12-month PFS will be evaluated by univariate analysis but different criteria for determination of PFS will be compared.
Compare the 12-month progression-free survival (PFS) of subjects receiving personalized or standard injected activity PRRT with ITMO criteria. | 12 months
  PFS will be determined by biochemical criteria (ITMO) on serial CT, and analysed independently. The 12-month PFS will be evaluated by univariate analysis but different criteria for determination of PFS will be compared.
Compare the 12-month progression-free survival (PFS) of subjects receiving personalized or standard injected activity PRRT with Choi criteria. | 12 months
  PFS will be determined by Choi criteria on serial CT, and analysed independently. The 12-month PFS will be evaluated by univariate analysis but different criteria for determination of PFS will be compared.

SECONDARY OUTCOMES:
Determine response rate of both treatment arms with RECIST1.1 criteria | 4 months
  Response rate as determined by structural criteria RECIST1.1
Determine response rate of both treatment arms with Choi criteria | 4 months
  Response rate as determined by structural criteria Choi.
Determine response rate of both treatment arms with ITMO criteria | 4 months
  Response rate as determined by structural criteria biochemical markers (ITMO criteria) (chromogranin A, 24h urinary HIAA).
Quality of life (QoL) questionnaire scores (EORTC QLQ30) will be compared between the two treatment arms | 8 months
  For QoL questionnaire scores (EORTC QLQ30) before, during, and after treatment
Quality of life (QoL) questionnaire scores (EORTC GINET21) will be compared between the two treatment arms | 8 months
  For QoL questionnaire scores (EORTC GINET21) before, during, and after treatment
Quality of life (QoL) questionnaire scores (EQ-5D) will be compared between the two treatment arms | 8 months
  For QoL questionnaire scores (EQ-5D) before, during, and after treatment
Correlation of QoL scores (EORTC QLQ30) to ctDNA | 8 months
  To assess correlation of QoL scores (EORTC QLQ30) to ctDNA allele frequency change from pre-treatment to on-treatment, using spearman correlation
Correlation of QoL scores (EORTC GINET21) to ctDNA | 8 months
  To assess correlation of QoL scores (EORTC GINET21) to ctDNA allele frequency change from pre-treatment to on-treatment, using spearman correlation
Correlation of QoL scores (EQ-5D) to ctDNA | 8 months
  To assess correlation of QoL scores (EQ-5D) to ctDNA allele frequency change from pre-treatment to on-treatment, using spearman correlation

OTHER OUTCOMES:
PFS and QoL scores to ctDNA levels | 8 months
  To assess correlation of PFS and QoL scores (EORTC QLQ30) to ctDNA levels (ctDNA allele frequency change from pre-treatment to on-treatment), the following tests will be used, Spearman correlation for quality of life and Kaplan- Meier curves stratified at a median for PFS.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Benard, MD, Principal Investigator — BC Cancer
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No